CLINICAL TRIAL: NCT05516173
Title: Role of Depression in Blood Pressure Control. A Cross-sectional Multicentric Study
Brief Title: Role of Depression in Blood Pressure Control. Study
Acronym: TUN-BP-BLUE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: General Administration of Military Health, Tunisia (Network)
Responsible Party: Sponsor
Other Study IDs: santémilitaire10
Record Dates: First submitted 2022-08-23; First posted 2022-08-25 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Hypertension; Depression
Keywords: Patient Health Questionnaire; Blood Pressure Monitoring, Ambulatory; hypertension; depression
MeSH Terms: conditions — Hypertension; Depression | interventions — Blood Pressure Monitoring, Ambulatory

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ambulatory patients: Patient with a high blood pressure during regular visit will undertake an ambulatory blood pressure monitoring. Before wearing the device , they will be asked to answer to the questionnaire and the investigators will gather their demographic,clinical characteristics and dietary habits data.
  Ethical considerations will be undertaken and respected.
  Interventions: Diagnostic Test: Blood Pressure Monitoring, Ambulatory

INTERVENTIONS:
Diagnostic Test: Blood Pressure Monitoring, Ambulatory — To monitor the blood pressure during 24 hours.

SUMMARY:
Our study aims to evaluate the role of depression in blood pressure control in ambulatory hypertensive patients.

DETAILED DESCRIPTION:
Research Problem: Hypertension is a multifactorial disease that affects approximately one quarter of the adult population. It is a major risk factor for stroke and cardiovascular disease.

Environmental and psychosocial factors play an important role in hypertension onset and control. The prevalence of depression among hypertensive patients is 26, 8% and its presence is associated with increased risk of cardiovascular-related morbi-mortality. Our study aims to evaluate the role of depression in blood pressure control in ambulatory hypertensive patients. Investigative process: This study is a cross-sectional, multicentric and descriptive study. the investigators intend to include three hundred and two patients. After obtaining their consent, a 24 hour ambulatory blood pressure monitor will be used to evaluate blood pressure control.

Depression was assessed by the 9-item-Patient Health Questionnaire (PHQ-9) in Tunisian dialect. Clinical, socio-environmental, psychosocial and therapeutic and prognosis data will be collected from medical records.

ELIGIBILITY:
Inclusion Criteria:

* Patients consulting for high blood pressure
* Patients older than 18 years.
* Patients able to give informed consent.

Non inclusion Criteria :

* Patients followed for depression under treatment.
* Hospitalized patients

Exclusion Criteria:

* a white coat hypertension

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: outpatients consulting in the cardiology department in the different participating centers .
Sampling Method: Non-Probability Sample
Enrollment: 302 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2022-11-15 (Estimated); Study Completion 2023-01-15 (Estimated)

PRIMARY OUTCOMES:
prevalence of depression in uncontrolled hypertensive patients. | on inclusion
  The prevalence of depression evaluated by PHQ9 in Tunisian dialect in hypertensive patients with abnormal ambulatory 24 hours blood pressure monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Aymen NOAMEN, MD, Principal Investigator — Military Hospital of Tunis; Wafa Fehri, Pr, Study Chair — Military Hospital of Tunis; Lilia Zakhama, Pr, Study Director — interior security forces hospital
Locations (4):
- Tunisia (4):
  - Interior Security Forces Hospital, La Marsa, Tunis Governorate
  - Regional hospital of Ben Arous, Ben Arous
  - Tahar Sfar regional hospital of Mahdia, Mahdia
  - Military Hospital of Tunis, Tunis

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Li Z, Li Y, Chen L, Chen P, Hu Y. Prevalence of Depression in Patients With Hypertension: A Systematic Review and Meta-Analysis. Medicine (Baltimore). 2015 Aug;94(31):e1317. doi: 10.1097/MD.0000000000001317. PMID 26252317
- [Derived] Raddaoui Y, Ben Amara A, Noamen A, Antit S, Hajri Y, Habli J, Ibn Hadj Amor H, Ben Youssef Y, Zakhama L, Fehri W. Role of depression in blood pressure control. A cross-sectional multicentric study. Tunis Med. 2024 Jan 5;102(1):7-12. doi: 10.62438/tunismed.v102i1.4723. French. PMID 38545723